CLINICAL TRIAL: NCT00036413
Title: A 12-week, Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicenter, Safety and Dose-ranging Study of Three Oral Doses (0.5 mg, 2.5 mg and 10 mg Once Daily) of TCH346 in Patients With Amyotrophic Lateral Sclerosis.
Brief Title: A 12-week, Multicenter, Safety and Dose-ranging Study of 3 Oral Doses of TCH346 in Patients With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTCH346 0102
Record Dates: First submitted 2002-05-09; First posted 2002-05-10 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — dibenzo(b,f)oxepin-10-ylmethyl-methyl-prop-2-ynyl-amine

INTERVENTIONS:
Drug: TCH346

SUMMARY:
This study is the first to be performed in Amyotrophic Lateral Sclerosis (ALS) patients with the novel compound TCH346. Its purpose is to evaluate the safety and clinical effects of 3 dose levels of TCH 346 compared to placebo in patients with a clinical diagnosis of laboratory-supported probable, probable or definite ALS. The study will require patients to visit the study center a total of at least 7 times over the course of up to 14 weeks. The study consists of 2 phases: A screening phase (up to 2 weeks) when patients will be evaluated for eligibility to participate in the study, and a double-blind treatment phase (12 weeks) when patients will receive daily doses of either TCH346 or placebo and will be evaluated for clinical effects. In addition, patients eligible to participate in this study will be required to have 3 magnetic resonance spectroscopic (MRS) scans. The MRS is a non-invasive, painless, "brain scan". The MRS will require traveling to a designated center in Montreal, Canada, which is very experienced in performing such MRS scans in ALS patients.

ELIGIBILITY:
* clinical diagnosis of laboratory-supported probable, probable, or definite ALS;
* have sporadic or familial ALS;
* have shown ALS symptom onset for no more than 3 yrs., inclusive, prior to randomization;
* FVC of >60%;
* ability to tolerate MRS evaluation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-01; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Safety of three oral doses of TCH346 versus placebo administered for up to 12 weeks to patients with ALS

SECONDARY OUTCOMES:
Biomarker assessments at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Neurological Institute, New York, New York, United States